CLINICAL TRIAL: NCT05157828
Title: A Cross-sectional Prospective Study of the Prevalence of Iron Deficiency Anaemia in Pregnant Patients Presenting for Antenatal Care at a Secondary Level Institution, Mowbray Maternity Hospital
Brief Title: Iron Deficiency Anaemia in Pregnant Patients Presenting for Antenatal Care
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Christella Alphonsus, Principal investigator, University of Cape Town
Other Study IDs: UCape Town
Record Dates: First submitted 2021-11-29; First posted 2021-12-15 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Iron Deficiency Anemia of Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a cross-sectional, prospective study of iron deficiency anaemia among pregnant patients presenting for antenatal care at a secondary level institution in the Western Cape, Mowbray Maternity Hospital, over a one-week period.

ELIGIBILITY:
Inclusion Criteria:

* All women presenting to the antenatal care services at Mowbray Maternity Hospital over the period of study recruitment.
* ≥ 18 years of age.
* Screen as anaemic (World Health Organisation <11g/dl) on bedside finger-prick haemoglobin.
* Who consent to participate.

Exclusion Criteria:

Patients who refuse to participate, and those under the age of 18 years will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients
Study Population: This study will include all consenting patients presenting to the Antenatal Clinic at Mowbray Maternity Hospital, for antenatal care, during the one-week period of recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of anaemia among all women presenting for antenatal care at a secondary level institution in the Western Cape, Mowbray Maternity Hospital, during a one-week period. | One week
  Proportion

CONTACTS AND LOCATIONS:
Overall Officials: Christella Alphonsus, MBChB, Principal Investigator — University of Cape Town
Locations (1):
- Mowbray maternity hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared by PI
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Not limoited
Access Criteria: Contact PI